CLINICAL TRIAL: NCT04016948
Title: A Multicenter Randomized Study of Real-time In-vivo Confocal Laser Endomicroscopy Optical Biopsy for Distal Margin in Low Rectal Cancer Compared to Intraoperative Frozen Section
Brief Title: Optical Biopsy for Distal Margin in Low Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Southern Medical University, China (Other); Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: yanjun
Record Dates: First submitted 2017-07-26; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; distal margin; confocal laser endomicroscopy; real-time; in vivo; optical biopsy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probe-based confocal laser endomicroscopy(pCLE) (Experimental): Confocal laser endomicroscopy optical biopsy will be performed in surgery for patients assigned to this group
  Interventions: Device: Probe-based confocal laser endomicroscopy optical biopsy
- Intra-operative frozen section(IFS) (Active Comparator): Intra-operative frozen section will be performed for patients assigned to this group
  Interventions: Device: Intra-operative frozen section

INTERVENTIONS:
Device: Probe-based confocal laser endomicroscopy optical biopsy — In the pCLE group, after intravenous injection of fluorescein, the optical biopsy will be performed, using a confocal miniprobe, to exam the rectal mucosa when the rectum transection is ready. The raters will analyse the CLE images to determine whether the distal margin is positive. In the IFS group, intra-operative frozen section will be performed at the site of distal margin after the rectum transection.
  Arms: Probe-based confocal laser endomicroscopy(pCLE)
Device: Intra-operative frozen section — In the pCLE group, after intravenous injection of fluorescein, the optical biopsy will be performed, using a confocal miniprobe, to exam the rectal mucosa when the rectum transection is ready. The raters will analyse the CLE images to determine whether the distal margin is positive. In the IFS group, intra-operative frozen section will be performed at the site of distal margin after the rectum transection.
  Arms: Intra-operative frozen section(IFS)

SUMMARY:
This is a multi-center prospective randomized controlled study. In this study, the investigators will use confocal laser endomicroscopy to make real-time in vivo optical biopsy of distal margin in rectal cancer surgery and help surgeons to make surgical decision.The investigators also assess the accuracy of CLE optical biopsy, compared with intra-operative frozen section.

DETAILED DESCRIPTION:
In low rectal cancer surgery, how to select the precise dissection plane and optimal surgical procedure is an important challenge for surgeons. In current clinic, surgeons select dissection plane by a comprehensive judgment of pre-operative pelvis MRI, colonoscopy and digital rectal examination, then through submitting the "doughnut" after cutting and anastomosis to intra-operative frozen section (IFS) to definite whether there is residual tumor in distal margin (DM). However, IFS can only make diagnosis using the tissue specimen in vitro and time-consuming. Once the IFS confirm positive margin, it always means anal resection should be implemented to ensure radical treatment. Therefore, if there is a real-time in situ examination method to evaluate DM in vivo, it will bring great benefits to both surgeons and patients.

Confocal laser endomicroscopy (CLE) had been widely used in medical field to diagnose colorectal disease, but it is seldom applied in surgical filed especially in rectal cancer to make optical biopsy and help surgical decision-making. Therefore, the investigators hypothesize that CLE can real-time in situ evaluate DM during surgery in rectal cancer and its accuracy is non-inferior to intra-operative frozen section.

In this study, the investigators will randomly assign patients to the experimental group (CLE optical biopsy) and control group (IFS). Using H-E staining pathological diagnosis as golden standard, the accuracy, sensitivity and specificity of both CLE optical biopsy and IFS will be evaluated and compared. And the investigators will also evaluate patients' postoperative urinary function, defection function and quality of life through a year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Ages from 18 to 70 years.
* Rectal tumor confirmed pathologically by endoscopic biopsy.
* The distance from lower edge of tumor to the dentate line is less than 5cm.
* Plan to perform curative resection.
* ASA(American Society of Anesthesiology)score class I,II,or III.
* Able to provide written informed consent.

Exclusion Criteria:

* Intestinal perforation or acute intestinal obstruction.
* Multiple distant metastasis and can not R0 resection.
* T4b according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition.
* Pregnancy or breastfeeding.
* Impaired renal function
* American Society of Anesthesiology score (ASA) class IV or V.
* Unable or refuse to provide written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of optical biopsy | One week after surgery
  Accuracy of confocal laser endomicroscopy optical biopsy of distal margin is determined by the pathology result.

SECONDARY OUTCOMES:
Sensitivity and Specificity | One week after surgery
  Sensitivity and specificity of confocal laser endomicroscopy optical biopsy of distal margin are determined by the pathology result.
Operation related indexes | One week after surgery
  Operation time in minutes
Postoperative function recovery | Up to 12 months
  Defecation and sphincter function will be combined to report Wexner score.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yan, M.D., Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rullier E, Laurent C, Bretagnol F, Rullier A, Vendrely V, Zerbib F. Sphincter-saving resection for all rectal carcinomas: the end of the 2-cm distal rule. Ann Surg. 2005 Mar;241(3):465-9. doi: 10.1097/01.sla.0000154551.06768.e1. PMID 15729069
- [Background] Gomes RM, Bhandare M, Desouza A, Bal M, Saklani AP. Role of intraoperative frozen section for assessing distal resection margin after anterior resection. Int J Colorectal Dis. 2015 Aug;30(8):1081-9. doi: 10.1007/s00384-015-2244-4. Epub 2015 May 16. PMID 25982468
- [Background] Kiesslich R, Gossner L, Goetz M, Dahlmann A, Vieth M, Stolte M, Hoffman A, Jung M, Nafe B, Galle PR, Neurath MF. In vivo histology of Barrett's esophagus and associated neoplasia by confocal laser endomicroscopy. Clin Gastroenterol Hepatol. 2006 Aug;4(8):979-87. doi: 10.1016/j.cgh.2006.05.010. Epub 2006 Jul 13. PMID 16843068
- [Background] Pech O, Rabenstein T, Manner H, Petrone MC, Pohl J, Vieth M, Stolte M, Ell C. Confocal laser endomicroscopy for in vivo diagnosis of early squamous cell carcinoma in the esophagus. Clin Gastroenterol Hepatol. 2008 Jan;6(1):89-94. doi: 10.1016/j.cgh.2007.10.013. Epub 2007 Dec 11. PMID 18063417
- [Background] Li Z, Zuo XL, Yu T, Gu XM, Zhou CJ, Li CQ, Ji R, Li YQ. Confocal laser endomicroscopy for in vivo detection of gastric intestinal metaplasia: a randomized controlled trial. Endoscopy. 2014 Apr;46(4):282-90. doi: 10.1055/s-0033-1359215. Epub 2014 Jan 28. PMID 24473908
- [Background] Li WB, Zuo XL, Li CQ, Zuo F, Gu XM, Yu T, Chu CL, Zhang TG, Li YQ. Diagnostic value of confocal laser endomicroscopy for gastric superficial cancerous lesions. Gut. 2011 Mar;60(3):299-306. doi: 10.1136/gut.2010.223586. Epub 2010 Dec 30. PMID 21193460
- [Background] Xie XJ, Li CQ, Zuo XL, Yu T, Gu XM, Li Z, Ji R, Wang Q, Li YQ. Differentiation of colonic polyps by confocal laser endomicroscopy. Endoscopy. 2011 Feb;43(2):87-93. doi: 10.1055/s-0030-1255919. Epub 2010 Oct 29. PMID 21038291
- [Derived] Tan J, Ji HL, Hu YW, Li ZM, Zhuang BX, Deng HJ, Wang YN, Zheng JX, Jiang W, Yan J. Real-time in vivo distal margin selection using confocal laser endomicroscopy in transanal total mesorectal excision for rectal cancer. World J Gastrointest Surg. 2022 Dec 27;14(12):1375-1386. doi: 10.4240/wjgs.v14.i12.1375. PMID 36632126